CLINICAL TRIAL: NCT00220649
Title: Phase I Study to Determine the Safety, Maximum Tolerated Dose, and Efficacy of Biweekly Oxaliplatin (Eloxatin) in Combination With Gemcitabine, Irinotecan, and 5-FU/Leucovorin (G-Flie) in Patients With Metastatic Solid Tumors or Adenocarcinoma of the Exocrine Pancreas
Brief Title: Safety Study of Combination Chemotherapy in Patients With Metastatic Solid Tumors or Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 175-03; OX-03-049
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Pancreatic Neoplasms
Keywords: solid tumors or adenocarcinoma of the exocrine pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Irinotecan; Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine; irinotecan; leucovorin; 5-fluorouracil; oxaliplatin

SUMMARY:
The purpose of this trial is to determine the maximum tolerated dose and the dose-limiting toxicity of biweekly oxaliplatin in combination with fixed doses of irinotecan, 5-fluorouracil/leucovorin and gemcitabine in patients with metastatic solid tumors or adenocarcinoma of the pancreas.

DETAILED DESCRIPTION:
Pancreatic cancer is a major health problem in the United States and other developed nations. Approximately thirty thousand cases of adenocarcinoma of the exocrine pancreas are diagnosed in the United States each year. The majority of these tumors are unresectable at the time of diagnosis. Unresectable and metastatic pancreatic cancer is often resistant to treatment with response rates of less than 10% and median survival times of less than six months associated with single agent chemotherapy. As of July 2003, gemcitabine remains the standard of care palliative chemotherapy for patients with locally advanced or metastatic pancreatic cancer. This drug has modest clinical activity. In a phase III randomized controlled trial, 126 patients with advanced symptomatic pancreatic cancer were randomized to receive either gemcitabine 1000 mg/m2 weekly x 7 followed by a week of rest and then weekly x 3 every 4 weeks thereafter or fluorouracil 600 mg/m2 once weekly. The primary endpoint was a score of clinical benefit response (CBR) derived from a composite of pain, performance status, and weight. CBR was experienced by 24% of the gemcitabine treated patients compared with 5% of 5-FU treated patients. The median survival durations were 5.65 and 4.41 months for gemcitabine-treated and 5-FU-treated patients, respectively. The one year survival was 18% for patients treated with gemcitabine compared to 2% for patients treated with 5-FU. The effectiveness of gemcitabine may be improved by altering the standard infusion schedule to a fixed dose rate. Gemcitabine requires intracellular phosphorylation to form active di- and triphosphates, which is dose rate dependent. A phase II trial randomized patients to either receive gemcitabine 2200 mg/m2 over a standard 30 minute infusion or gemcitabine 1500 mg/m2 at a fixed rate of 10 mg/m2/min weekly x 3 every 4 weeks. The fixed rate infusion of 10 mg/m2/min was associated with a higher response rate of 16.6% v 2.7%, longer median survival 6.1 v 4.7 months, and a higher percentage of patients surviving one year or more, 23% v 0%. The fixed rate infusion schedule was also associated with significantly higher median gemcitabine triphosphate levels in peripheral circulating mononuclear cells after each infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of a solid tumor, OR advanced or metastatic disease that is refractory to conventional treatment or for which no standard therapy exists.
2. Age > 18 years old.
3. A performance status of ≥ 60 on the Karnofsky scale
4. Life expectancy of at least 12 weeks.
5. Patients must give written informed consent as per institutional and federal regulatory requirements.
6. No chemotherapy, immunotherapy or radiotherapy for at least four weeks prior to entry in the study (six weeks for nitrosureas or mitomycin C). Patients may not receive concurrent chemotherapy, immunotherapy or radiotherapy while participating in this study. Patients may not receive concurrent treatment with any other investigational drug while on this protocol.
7. Patients must have measurable or evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST).
8. Absolute granulocyte count of > 1,500/mm3 and a platelet count > 100,000/mm3.
9. Patients must have adequate liver and renal function defined by a bilirubin of ≤ 2.0 mg/dl, and a creatinine of ≤ 1.5 mg/dl respectively.
10. Patients must be able to stay in the general area for the duration of their treatment on this clinical research study.
11. Men and women who are fertile must use adequate contraception. Premenopausal women must have a negative pregnancy test documented prior to study entry.
12. Patients must be disease-free of prior invasive malignancies for >= 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.

Exclusion Criteria:

Individuals excluded from participating in this study are described below.

1. Women who are pregnant or breast-feeding
2. Patients with clinical signs of brain involvement or leptomeningeal disease.
3. Patients with progressive sensory neuropathy or progressive hearing loss or tinnitus.
4. Patients with other serious illness or medical conditions, including but not limited to the following:

   * congestive heart failure or angina pectoris
   * previous history of myocardial infarction within 1 year from study entry
   * uncontrolled hypertension or arrhythmias
   * active infections
   * unstable diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-03

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and the dose-limiting toxicity (DLT) of biweekly oxaliplatin in combination with fixed doses of irinotecan, 5-fluorouracil/leucovorin and gemcitabine

SECONDARY OUTCOMES:
To document any antitumor activity with biweekly oxaliplatin in combination with fixed doses of irinotecan, 5-fluorouracil/leucovorin and gemcitabine administered on this schedule

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kozuch, Principal Investigator — Continuum Cancer Center
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States